CLINICAL TRIAL: NCT06979713
Title: Yoga, Education, and Nidra (YEN) for Chronic Low Back Pain: A Pilot Study on Pain Modulation, Well-Being, and Sleep
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Responsible Party: Principal Investigator, Abigail Wilson, Assistant Professor, University of Central Florida
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11
Record Dates: First submitted 2025-05-13; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga, Pain Education, Yoga Nidra (Experimental): Yoga postures targeting lower back, pain education, yoga nidra with pain acceptance intention and motor imagery.
  Interventions: Other: yoga, pain education, yoga nidra
- Yoga, Pain Education, Relaxing Music (Active Comparator): Yoga postures targeting lower back, pain education, relaxing music
  Interventions: Other: yoga, pain education, relaxing music

INTERVENTIONS:
Other: yoga, pain education, yoga nidra — Participants will complete a series of yoga postures targeting the lower back combined with pain education. The session will conclude with either yoga nidra with pain acceptance intention. Interventions are completed at home 2x/week for 6 weeks.
  Arms: Yoga, Pain Education, Yoga Nidra
Other: yoga, pain education, relaxing music — Participants will complete a series of yoga postures targeting the lower back combined with pain education. The session will conclude with relaxing music depending on group assignment. Interventions are completed at home 2x/week for 6 weeks.
  Arms: Yoga, Pain Education, Relaxing Music

SUMMARY:
The purpose of this study is to compare the impact of yoga, pain education, and yoga nidra with pain acceptance intention to yoga, pain education, and relaxing music on pain intensity, well-being, and sleep quality. This is a pilot study trial of individuals with chronic low back pain. Participants will attend two sessions in the laboratory (week 1 and week 8) and complete their assigned intervention 2 x per week for 6 weeks at home. Participants will be randomized to either receive yoga postures targeting the low back, pain education, and yoga nidra with pain acceptance intention and motor imagery or yoga postures targeting the low back, pain education, and relaxing music.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain in lower back that has lasted for over three months
* Pain intensity rated as 3/10 or higher in the past 24 hours (0=no pain, 10=worst pain imaginable)

Exclusion Criteria:

* non-English speaking
* systemic medical conditions that affect sensation (such as uncontrolled diabetes)
* History of surgery or fracture within the past six months
* any blood clotting disorders (such as hemophilia)
* any contraindication to the application of ice (blood pressure > 140/90 mmHg, cold urticaria, cryoglobulinemia, paroxysmal cold hemoglobinuria, circulatory compromise)
* Exceed pressure and heat sensory thresholds
* Unable to access the internet or email
* Pregnant
* Unable to exercise without medical clearance (assessed on PAR-Q+ on first visit)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | Completed on week one and week eight
  Participants will rate their low back pain from 0=no pain to 100=worst pain imaginable.
Warwick-Edinburgh Mental Well-Being Scale | Completed on week one and week eight
  Self-report measure of well-being
Pittsburgh Sleep Quality Index | Completed on week one and week eight
  Self-report measure of sleep quality

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No